CLINICAL TRIAL: NCT04132674
Title: Switching to a Fixed Dose Combination of Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF) in HIV-1 Infected Marginalized Populations Who Are Virologically Suppressed
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver Infectious Diseases Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Biktarvy Study
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Human Immunodeficiency Virus I Infection; Drug Use
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- B/F/TAF (Other): Switching participants who are currently on multi-tablet HIV antiretroviral therapy, including multi-tablet regimens and/or two drug combinations (dual therapy) to one oral tablet of B/F/TAF once-daily for 72 weeks
  Interventions: Drug: Bictegravir/emtricitabine/tenofovir alafenamide

INTERVENTIONS:
Drug: Bictegravir/emtricitabine/tenofovir alafenamide — Taking one oral tablet of B/F/TAF once-daily for 72 weeks

SUMMARY:
In an effort to engage more HIV-infected PWUD into care, and ensure treatment adherence and efficacy, simplification of older, multi-tablet regimens is required. Newer, more potent molecules can also overcome resistant that has persisted with previous regimens, while simultaneously providing a high barrier to resistance. The co-formulation of B/F/TAF is a viable switch-option for patients who have experienced lower adherence with previous regimens due to high pill burden, or for those requiring a more potent regimen due to emergent resistances. The formal evaluation of B/F/TAF in this context will allow us to optimize care for HIV-infected PWUD.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥19 years of age infected with HIV-1
2. Participant has an undetectable viral load <40 copies/mL at screening with any CD4 count and has exhibited any, or all of the following:

   1. Transient HIV viremia (episodes of HIV viral load between 40-1000 copies/mL) in the past 12 months, OR Virologic breakthrough (HIV viral load > 1000 copies/mL) in the past 12 months, OR Documented instances of non-adherence for a period of more than 7 days or…
   2. Participant is currently on multi-tablet HIV antiretroviral therapy, including multi-tablet regimens and/or two drug combinations (dual therapy)
   3. Participant has a history or current indication of illicit drug use.
   4. Patients infected with HCV and or HBV can be included in this study.
   5. If female, participant must have a negative pregnancy test and agree to use, for the duration of the study, a method of birth control that has a history of proven reliability as judged by the investigator.

Exclusion Criteria:

1. They have any documented history of integrase inhibitor resistance
2. They exhibit any of the following:

   1. Creatinine Clearance Rate < 30 ml/min
   2. Hemoglobin < 10.0 g/dL
   3. Absolute neutrophil count <750 cells/mL
   4. Platelet count < 50,000 /mL
   5. ALT or AST >5x upper limit of normal (ULN)
   6. Creatinine > 1.5x ULN
3. They are taking medication that is contraindicated with any component of B/F/TAF.
4. They are pregnant or breastfeeding.
5. They do not/have not ever used any form of illicit drug use.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects that remain virally suppressed at week 48 | Interim analysis of efficacy will be done at 24 weeks
  The proportion of subjects with HIV RNA <40 copies/mL

SECONDARY OUTCOMES:
The proportion of subjects with viral blips | Analysis will be done at 72 weeks
  Viral blips defined as detectable HIV viral load between 40-1000 copies/mL at week 72
Changes of adherence | Analysis will be done at 72 weeks
  Changes of adherence from baseline at week 2, 8, 24, 48, and 72 with an adherence questionnaire
Proportion of patients that achieved >90% adherence | Analysis will be done at 72 weeks
  Proportion of patients that achieved >90% adherence
The proportion of viral blips on regimens pre-switch compared to the blips on B/F/TAF | Analysis will be done at 72 weeks
  The proportion of viral blips on regimens pre-switch compared to the blips on B/F/TAF
The proportion of participants that discontinued B/F/TAF due to side-effects at weeks 36 and72 | Analysis will be done at 72 weeks
  The proportion of participants that discontinued B/F/TAF due to side-effects at weeks 36 and72
Changes to baseline quality of life at week 4, 12, 36, 60, and 72 using the HIV Symptoms Distress Module | Analysis will be done at 72 weeks
  Changes to baseline quality of life at week 4, 12, 36, 60, and 72 using the HIV Symptoms Distress Module

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Vancouver Infectious Diseases Centre, Vancouver, British Columbia
  - Victoria Cool Aid Society, Victoria, British Columbia